CLINICAL TRIAL: NCT06596941
Title: Ultrasound Assessment of Isolated Distal Deep Vein Thrombosis
Acronym: IDDVT
Status: Active, not recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MR-31-24-020092
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Iddvt; Pulmonary Embolism (PE)
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Retrospective assessment of ultrasound and clinical characteristics of patients with IDDVT, development of a pulmonary embolism risk prediction model for thrombus, and provision of appropriate diagnostic and therapeutic recommendations.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of new-onset IDDVT confirmed by lower limb vascular ultrasound; presence/absence of pulmonary embolism clarified by pulmonary artery CTA; ultrasound and pulmonary artery CTA results spanning no more than 5 days.

Exclusion Criteria:

Anticoagulation therapy in the last month; pregnancy or puerperium; recurrent DVT or PE.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Both male and female
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
IDDVT with PE | At the initial visit
  IDDVT patients with concomitant PE

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No